CLINICAL TRIAL: NCT02523144
Title: A Qualitative Comparison of Oral Chloral Hydrate vs 2.0 or 3.0 mcg/kg Nasal Dexmedetomidine in Children Undergoing Transthoracic Echocardiography
Brief Title: Dexmedetomidine in Children Having Transthoracic Echocardiography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCMCIRB-K2014057
Record Dates: First submitted 2015-07-27; First posted 2015-08-14 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Heart Disease
Keywords: Transthoracic echocardiography; echo; TTE
MeSH Terms: conditions — Heart Diseases | interventions — Chloral Hydrate; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chloral Hydrate + placebo (Active Comparator): Oral chloral hydrate sedation in flavored syrup plus nasal saline placebo
  Interventions: Drug: Chloral Hydrate; Drug: Placebo
- Dexmedetomidine 2mcg/kg + placebo (Active Comparator): Nasal dexmedetomidine sedation 2 mcg/kg plus oral flavored syrup placebo
  Interventions: Drug: Dexmedetomidine; Drug: Placebo
- Dexmedetomidine 3mcg/kg + placebo (Active Comparator): Nasal dexmedetomidine sedation 3 mcg/kg plus oral flavored syrup placebo
  Interventions: Drug: Dexmedetomidine; Drug: Placebo

INTERVENTIONS:
Drug: Chloral Hydrate — 70mg/kg chloral hydrate
  Arms: Chloral Hydrate + placebo
Drug: Dexmedetomidine — 2mcg/kg
  Arms: Dexmedetomidine 2mcg/kg + placebo
Drug: Dexmedetomidine — 3mcg/kg
  Arms: Dexmedetomidine 3mcg/kg + placebo
Drug: Placebo — Flavored placebo syrup

SUMMARY:
Sedation Techniques for children undergoing transthoracic echocardiography (TTE).

DETAILED DESCRIPTION:
The goal in this study is to determine if there is a significant difference in the quality of sedation between two standard sedation techniques and between two doses of dexmedetomidine for children undergoing (TTE).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients scheduled to receive sedation for transthoracic echocardiography
* Subject must be a candidate for both types of anesthetic and both doses of dexmedetomidine
* Must be 3 months to 36 months of age

Exclusion Criteria:

* The subject has a history of cardiac conduction system disease (e.g. 1st or 2nd degree AV block) or channelopathy (e.g. long QT).
* The subject is taking digoxin, alpha-adrenergic or beta-adrenergic agonist or antagonist (e.g., clonidine, propranolol, albuterol), anti-arrhythmic medications, or vasodilators (e.g. ACE inhibitors)
* The subject has received a dose of any other sedative within 48 hours.
* The subject has life-threatening, medical conditions (American Society of Anesthesiologists Physical Status 4, 5). The American Society of Anesthesiologists (ASA) classification scale is a measure of physical status or how healthy the patient is. For our study, we will focus on children which are defined as ASA I, II or III which means a healthy child (ASA I), a child with a systemic disease that is mild and well controlled (ASA II) or a child with systemic disease that is severe and controlled (ASA III).
* The subject is allergic to or has a contraindication to any of the drugs used in the study.
* The subject has previously been treated under this protocol.
* The subject has severe coarctation of the aorta (risk of exaggerated vasoconstriction)
* The subject has Moyamoya disease (risk of recurrent stroke)

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 279 (Actual)
Dates: Start 2014-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Time to sedation | 30 minutes
  Achieve Ramsay sedation >3 within 30 minutes of administration of drug

SECONDARY OUTCOMES:
Duration of sedation level >3 | Patients will be followed for the duration of the procedure, average of 1 hour
The number of sonographer pauses | Participants will be followed for the duration of the procedure, average of 1 hour
  The number of sonographer pauses over 2 minutes due to patient movement or medical interventions will be counted
Need for rescue dexmedetomidine | Participants will be followed for the duration of the procedure, average of 1 hour
  The incidence of need for rescue nasal dexmedetomidine, due to patient arousal or movement prior to completion of TTE.
Incidence of respiratory complications | Participants will be followed for the duration of the hospital stay, average of 2 hours
  Documentation of the incidence of respiratory complications
Vital sign deviations of more than 30% from baseline | Participants will be followed for the duration of the hospital stay, average of 2 hours
  Documentation of the incidence of blood pressure or heart rate deviations of more than 30% from baseline. Baseline will be measured prior to sedative administration.
Post anesthesia drowsiness | Participants will be followed for the duration of the post procedure stay, average of 1 hour
  Documentation of the incidence of post anesthesia drowsiness
Duration of Post Anesthesia Care Unit phase | Participants will be followed for the duration of the post procedure stay, average of 1 hour
  Documentation of the stay in Post Anesthesia Care Unit in minutes
Time to oral fluid intake | Participants will be followed for the duration of the post procedure stay, average of 1 hour
  Documentation of the time (in minutes) to oral fluid intake during the PACU phase
Time to discharge | Participants will be followed for the duration of the post procedure stay, average of 1 hour
  Documentation of the hospital stay after completion of the TTE.
Satisfaction of parents | Up to 3 days
  The satisfaction of the sedation technique will be completed by the parents by asking a series of questions during a follow-up phone call the next business day after the TTE.
Severity of respiratory complications | Participants will be followed for the duration of the hospital stay, average of 2 hours
  Documentation of the severity of respiratory complications
Post anesthesia agitation | Participants will be followed for the duration of the post procedure stay, average of 1 hour
  Documentation of the incidence of post anesthesia agitation

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miller, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Shanghai Children's Hospital, Shanghai, China